CLINICAL TRIAL: NCT07352748
Title: Exploiting Heterogeneity in Hormone Therapy Response to Reveal Early Determinants of Drug Resistance in Advanced PCa
Acronym: MOSAIC
Status: Active, not recruiting | Type: Observational
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Francesca Zacchi, Medical Doctor, Universita di Verona
Other Study IDs: 296CET
Record Dates: First submitted 2025-09-23; First posted 2026-01-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with histological diagnosis of advanced prostate cancer who started hormone therapy: A fresh tumor biopsies and FFPE block will be taken at baseline and after 4 weeks of hormone therapy and/or AR targeting agents. Blood samples for the isolation of plasma, serum and PBMC will be collected before the start of therapy and after 4 weeks of hormone therapy and/or AR targeting agents. The correlation of biopsies analyses and clinical data will advance the understanding of prostate cancer progression pathways and guide the design of subsequent studies in the field of personalized medicine.
  Interventions: Procedure: biopsy
- Patients due for prostate biopsy to confirm the diagnosis of a prostate adenocarcinoma at high risk: A fresh tumor biopsies and FFPE block and blood samples for the isolation of plasma, serum and PBMC will be taken at baseline. This cohort was necessary because it is complex to intercept patients at the time they perform diagnostic biopsy and then obtain fresh biopsies pre-hormonal treatment. If patients of this group will metastasize, these patients will be incorpored in the other.
  Interventions: Procedure: Prostate biopsy

INTERVENTIONS:
Procedure: biopsy — A fresh tumor biopsies and an FFPE block will be taken at baseline (alternatively, as a basal biopsy could be used archival FFPE tumor material left over from surgical procedures or previous biopsies if available and if a fresh biopsy at baseline is not feasible or safe; in case of availability of frozen and FFPE archival blocks, 1 frozen block and 1 FFPE block will be used for the analyses) and after 2-4 weeks of hormonal treatment with ADT and/or AR inhibitors. Biopsies will be performed guided by ultrasound or CT, depending on location. From each Fresh biopsy, 2 core biopsies will be collected, 1 will be processed into an FFPE block, and the second will be processed according to freezing procedures.
  Groups: Patients with histological diagnosis of advanced prostate cancer who started hormone therapy
Procedure: Prostate biopsy — Fresh and FFPE block tumor biopsies at baseline
  Groups: Patients due for prostate biopsy to confirm the diagnosis of a prostate adenocarcinoma at high risk

SUMMARY:
The goal of this observational study is to study intra-patient tumor and TME heterogeneity after initiation of hormonal therapy (ADT +- ARSI), while the patient is responding to treatment, to understand the drivers of hormonal therapy resistance and identify potential novel therapeutic targets in metastatic prostate cancer patients. The main question it aims to answer if intra-tumor adaptive mechanisms including expression of immune checkpoint proteins and changes in the tumor immune infiltrate are related to the induction of a senescent phenotype in response to hormonal therapy.

Participants will asked to provide an FFPE and/or fresh biopsy sample from the primary tumor or a metastatic site at baseline (before starting hormonal therapy) and during the course of hormonal therapy. Additionally, a maximum of 2 blood tubes (10ml) will be collected each time.

ELIGIBILITY:
Inclusion Criteria Group A:

* Patients with histological diagnosis of advanced prostate cancer (defined as the presence of metastatic disease, including both metastatic hormone naïve prostate cancer patients and metastatic castration resistant prostate cancer patients);
* Patients who started ADT or ADT plus AR inhibitor therapy (Enzalutamide, Darolutamide or Apalutamide or Abiraterone) in a standard therapy.
* Have accessible metastatic and/or primitive disease to perform a biopsy safely during hormonal therapy (ADT or ADT plus AR inhibitor therapy) and before hormonal therapy (alternatively, as a basal biopsy could be used archival FFPE or frozen tumor material left over from surgical procedures or previous biopsies, if available)
* Written acceptance of informed consent to be included in the present study.
* Aged 18 or over.

Inclusion Criteria Group B:

* Patients due for prostate biopsy to confirm the diagnosis of a prostate adenocarcinoma at high risk of metastatic disease. High risk is defined as follows:
* PSA >=20ng/dL with or without imaging suggestive of metastatic prostate cancer OR
* PSA >=10 ng/mL and <= 20 ng/mL AND >=33% risk to have a high grade disease on prostate biopsy according to the MSKCC nomogram "Risk of high grade cancer of prostate biopsy" (https://www.mskcc.org/nomograms/prostate/biopsy_risk_dynamic).
* Written acceptance of informed consent to be included in the present study.
* Aged 18 or over

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer receiving care at Azienda Ospedaliera Universitaria Integrata di Verona, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2026-10-17 (Estimated)

PRIMARY OUTCOMES:
A) Density of tumor-infiltrating immune cells | From enrollment to 24 months
  Description: Density of tumor-infiltrating lymphocytes (CD3+, CD4+, CD8+, FOXP3+) assessed by multiplex immunohistochemistry in tumor biopsies from patients under hormonal therapy.
  Unit of Measure: Cells/mm²
Tumor expression of Immune checkpoints | From enrollment to 24 months
  The investigators will pursue IHC assessment of immunomodulatory proteins. I will use a multiplexed customized IHC panel and the expression of the immunomodulatory proteins will be assessed in a semiquantitative manner (negative, 1+, 2+, 3+) in different tumor areas. I will compare the expression of immunomodulatory proteins assessed on human prostate cancer biopsies under hormonal treatment with same-patient pre-treatment therapy biopsies.
Emergence of a senescent phenotype | From enrollment to 24 months
  The investigators will confirm in vivo, in human samples, the senescent phenotype described in prostate cancer preclinical models, assessing the SA-Beta-Gal activity on fresh OCT-embedded biopsies and/or testing the telomere shortening in FFPE biopsies, depending If will be feasible to collect both fresh frozen and FFPE cores biopsies.
Changes in expression of prostate cancer-specific markers and therapeutic targets. | From enrollment to 24 months
  The investigators will also test the expression of prostate cancer specific markers PSMA, STEAP1, STEAP2 in response to AR blockade by IHC in pre-treatment vs post-treatment samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Verona, Verona, VR, Italy